CLINICAL TRIAL: NCT01923038
Title: Re-expansion of Atelectasis During Laparoscopic Surgery. Recruitment Maneuver vs Positive End-expiratory Pressure: a Randomized Study
Brief Title: Evaluation of Ventilatory Strategies During Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Vittoria Hospital (Other)
Responsible Party: Principal Investigator, Emilpaolo Manno, Emergency Department Director, Maria Vittoria Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCB232; MariaVittoria Hospital (Other: MariaVittoria Hospital)
Record Dates: First submitted 2013-05-17; First posted 2013-08-14 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Pneumonia
Keywords: atelectasis; laparoscopic surgery; anesthesia; mechanical ventilation; Prevent; shape of the airway; pressure-time curve
MeSH Terms: conditions — Pneumonia; Pulmonary Atelectasis | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Patients ventilated with zero end expiratory pressure (ZEEP) (Active Comparator): patients undergoing gynecologic laparoscopic surgery ventilated at zero end expiratory pressure
  Interventions: Procedure: First arm: patients ventilated with zero end expiratory pressure
- Patients ventilated with positive end expiratory pressure (Active Comparator): patients undergoing gynecologic laparoscopic surgery ventilated at PEEP
  Interventions: Procedure: Patients ventilated with Positive End Expiratory Pressure
- recruitment plus PEEP (Active Comparator): patients undergoing gynecologic laparoscopic surgery undergoing recruitment plus PEEP
  Interventions: Procedure: Patients ventilated with Positive End Expiratory Pressure plus Recruitment maneuver

INTERVENTIONS:
Procedure: First arm: patients ventilated with zero end expiratory pressure
  Arms: Patients ventilated with zero end expiratory pressure (ZEEP)
Procedure: Patients ventilated with Positive End Expiratory Pressure
  Arms: Patients ventilated with positive end expiratory pressure
Procedure: Patients ventilated with Positive End Expiratory Pressure plus Recruitment maneuver
  Arms: recruitment plus PEEP

SUMMARY:
Atelectasis involving declive areas often occurs during general anesthesia and may persist postoperatively. This phenomenon could be amplified by pneumoperitoneum and Trendelenburg position. Hypothesis: To evaluate whether the shape of the airway pressure-time curve, Stress Index (SI), during constant flow inflation can lead ventilator setting during general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesiology (ASA) I, II;
* age > 18 years;
* elective surgery

Exclusion Criteria:

* ASA III, IV;
* Age < 18 years;
* emergency surgery

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pulmonary Stress Index | Continuous evaluation during time of surgery. Partecipants will be followed for the duration of hospital stay, an expected average of 1 weeks

SECONDARY OUTCOMES:
Cardiac Index | Continuous evaluation during the time of surgery

OTHER OUTCOMES:
Blood gases | Continuous evaluation during the time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Emilpaolo Manno, MD, Study Director — Maria Vittoria Hospital
Locations (1):
- Maria Vittoria Hospital, Turin, Turin, Italy